CLINICAL TRIAL: NCT02535702
Title: Development of Neuroimaging Methods to Assess the Neurobiology of Addiction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 150186; 15-AA-0186
Record Dates: First submitted 2015-08-28; First posted 2015-08-31 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-11-26

CONDITIONS: Normal Physiology
Keywords: fMRI; EEG

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Attentional Bias Task (Experimental): Subjects will briefly see two images side by side on a screen. Immediately after, a dot appears on the left or on the right. The subjects task is to press the left or right button, following the position of the image (left or right). Images can contain food-related items. We will also show short 1-minute food-related movies. Subjects will be asked to fast for three hours before this task begins.
  Interventions: Other: In vivo MRS; Other: fMRI; Other: Stimulation tasks
- Cue Reactivity Task (Experimental): In this task subjects will view pictures of various items on the screen in front of them. Subjects will rate the items by how much they would like to have them. Subjects will choose how much they want the item by pressing a button.
  Interventions: Other: In vivo MRS; Other: fMRI; Other: Stimulation tasks
- Delay Discounting Task (Experimental): Subjects will be asked to imagine whether they would receive money now or money later (in the future). The future money option may be several days from now or as far out as 6 weeks from now. For example, a s ubject may see a $100 option in 6 weeks or a $10 option now. Subjects will not receive actual money for participation in this task
  Interventions: Other: In vivo MRS; Other: fMRI; Other: Stimulation tasks
- Motivational Reward Task (Experimental): Subjects will make a choice among some items presented on the screen in front of them. One of the items will be the winner item. The other items will be loser items. Each time a subject is presented with various items, they will choose the item they think is the winner item. Subjects will start with bonus points at the beginning of the task, so they can add more points to this amount as they continue to choose winner items.
  Interventions: Other: In vivo MRS; Other: fMRI; Other: EEG/EOG; Other: Stimulation tasks
- NSPRD Task (Experimental): During the MRI scan, subjects will get small electric shocks through electrodes placed on one of their toes. The shocks feel like an elastic band snapping against the skin. Right after a shock, subjects will see a dot on the computer screen. Subejcts will press a button to rate the intensity of the shock.
  Interventions: Other: In vivo MRS; Other: fMRI; Other: NSPRD
- Reasoning Task (Experimental): Subjects will identify changes in various shapes when they are displayed on the screen in front of them. Some changes of the shapes may be that they were rotated, enlarged, or multiplied. Subjects will choose the changes in the shapes by pressing a button.
  Interventions: Other: In vivo MRS; Other: fMRI; Other: Stimulation tasks
- Respiratory Challenge (RC) Task (Experimental): Participants will be visually instructed to take a brief deep breath (inhale) and release the breath (exhale). They will inhale and exhale one more time with visual cues at specific times (60 seconds, 120 seconds, 180 seconds, 240 seconds, etc. with successive 60 seconds intervals). A black cross will remain centered on a grey slide during the normal respiration periods. To signal the RC periods, the slide will change color to yellow READY slide, then to green BREATHE IN slide, then to blue BREATHE OUT slide. The sequence will repeat one more time to Breath In and Breath Out and then finally go back to the yellow Breathe Normally slide. The instruction words will be written on the slides. Each slide will be shown for 3 seconds. The task will take a total of 15 minutes (total of 900 seconds with 14 RC periods).
  Interventions: Other: In vivo MRS; Other: fMRI; Other: Stimulation tasks; Other: Structural MRI
- Self-control Task (Experimental): During the MRI scan, subjects will do a task that requires close concentration. Subjects will be asked to respond quickly to images on the computer screen, during which they will hear distracting noises. The subject will be able to remove the distraction in order to complete the task. During some sub-study sessions, subjects will start with no money ($0) and may be able to earn up to $40 if they do not remove the distraction. At other sub-study sessions, subjects will start with $40 and may lose between 25 to $1 each time they remove the distraction. Subjects cannot lose more than $40 in these sessions. Compensation for this sub-study is up to $40 per session, depending on their performance.
  Interventions: Other: In vivo MRS; Other: fMRI; Other: Stimulation tasks
- Spinner Task and MID Task (monetary incentive delay task) (Experimental): The Spinner task requires the subject to participate in a game of chance while lying in the MRI scanner. Subjects will be asked to respond by pressing a button. The MID task is a reaction time task. The MID Task tests how quickly a subject can press a button to hit a target on the screen in front of them. If the subject presses the button as soon as the target appears, the subject will score points. Subjects should try to score as many points as you can.
  Interventions: Other: In vivo MRS; Other: fMRI; Other: Stimulation tasks

INTERVENTIONS:
Other: In vivo MRS — 1H MR spectroscopy to assess brain metabolites.
Other: fMRI — Three fMRI sessions to assess test-retest reliability of functional connectivity (FC) measures at rest and during task performance.
Other: EEG/EOG — Electroencephalography or electrooculography (EEG/ EOG) sessions to record electrical activity of the brain or measure corneo-retinal standing potentials.
  Arms: Motivational Reward Task
Other: Stimulation tasks — To be used in the context of fMRI to study blood-oxygenation-level- dependent responses in the brain to sensory stimulation.
  Arms: Attentional Bias Task; Cue Reactivity Task; Delay Discounting Task; Motivational Reward Task; Reasoning Task; Respiratory Challenge (RC) Task; Self-control Task; Spinner Task and MID Task (monetary incentive delay task)
Other: NSPRD — To be used in conjunction with pupillometry in the context of fMRI to study blood-oxygenation-level-dependent responses to selective neurostimulation of pain fibers.
  Arms: NSPRD Task
Other: Structural MRI — High spatial MRI and diffusion tensor imaging (DTI) to assess brain morphology and structural connectivity.
  Arms: Respiratory Challenge (RC) Task

SUMMARY:
Background:

Abusing alcohol, drugs, and other substances can cause serious health problems. These substances also can affect brain function. Researchers want to learn more about brain function by using magnetic resonance imaging (MRI). This uses a magnetic field and radio waves to take pictures of the brain.

Objective:

To develop new ways to use MRI to study the brain.

Eligibility:

Healthy people 18 years of age or older.

Design:

Participants will be screened with a medical history, physical exam, and blood and urine tests.

They will answer questions about their drug use and psychiatric history. They will be asked about family history of alcoholism or drug abuse.

Participants will answer questions to see if they can participate in MRI.

Participants will have MRI scans. The scanner is a metal cylinder in a strong magnetic field. Participants will lie on a table that slides in and out of the cylinder. A device called a coil may be placed over the head.

Each sub-study will include up to 3 different MRI visits. Participants can be in multiple sub-studies. But they can have only 1 MRI per week and 20 per year.

During MRI visits, participants may have urine collected. They may get another MRI questionnaire.

Participants may have a clinical MRI brain scan. This may show physical problems in the brain.

During some scans, participants may perform simple movement, memory, and thinking tasks.

Participants may be connected to a machine to monitor brain activity during the scan. Small metal electrodes will be placed on the scalp. A gel will be placed in the space between the electrodes and the scalp.

...

DETAILED DESCRIPTION:
* Objectives: To improve sensitivity as well as spectral and spatiotemporal resolutions in magnetic resonance (MR) studies assessing structural, neurochemical, hemodynamic and electrophysiological changes that occur in the human brain during the resting state as well as those that occur in response to novel sensory, motor, cognitive or emotional stimulation paradigms.
* Study population: We intend to complete studies in 128 healthy volunteers, (64 males and 64 females, 18 years or older).
* Design: We will conduct pilot studies, each with up to 16 subjects, to optimize MR pulse sequences and/or functional MR imaging (fMRI) task paradigms pertinent to the theme of Addiction . MR pulse sequences and/or fMRI task paradigms will be validated against

appropriated gold-standard methods/tasks. These studies are required to maximize the sensitivity of new imaging techniques and fMRI tasks used for clinical and research applications that take advantage of 3T MRI scanners at NIH. If an exploratory study leads to results of interest, and if a larger population is necessary to reach statistical significance, a separate protocol will be submitted with a priori hypotheses, specific study design and power analysis adapted from the pilot studies performed in the present protocol.

* Outcome parameters: Although multiple measures will be collected, the primary outcome will be amplitude and reliability of regional-specific BOLD fMRI signals.
* MRI: we will analyze measures such as the amplitude and the reliability of the test-retest measures of fMRI signals; functional connectivity metrics; tractography between seed and target regions of interest (diffusion tensor imaging, DTI); brain morphometry (using

automatic segmentation and voxel-brain morphometry, VBM); and brain metabolite levels in regions of interest (using MR spectroscopy, MRS).

* EEG (electroencephalography): we will quantify measures such as event or task-related potentials, and coherence between sensors or sources located close to the brain areas of interest.
* Behavioral measures: during fMRI we will quantify measures such as reaction times and accuracy (using MRI compatible response pads) as well as eye movement (using MRI compatible eye trackers) and self-reports of the study experience (i.e., degree of interest

and motivation and alertness).

-Physiological measures: During fMRI, we will record physiological parameters such as blood pressure, skin conductance, respiratory frequency, or heart rate, to interpret outcome measures.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Eighteen years or older.
  2. Ability to provide written informed consent as determined by physical examination and verbal communication. Capacity to consent will be determined by those obtaining the informed consent.
  3. Willingness to abstain from drug use on scheduled testing days.

EXCLUSION CRITERIA

1. Positive urine pregnancy test in females.
2. Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head (including but not limited to pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments) or fear of enclosed spaces as determined by the self-report checklist.
3. Claustrophobia.
4. Body weight >550 lbs, which is the weight limit of the MR scanner.
5. Current DSM-5 diagnosis of a psychiatric disorder (other than nicotine/caffeine use disorders) as determined by history and clinical exam including substance use disorder, alcoholism and alcohol dependence. Past history of a mental disorder as defined by DSM-IV or DSM-5 will be excluded only if it was severe enough as to require hospitalization (any length), or chronic medication management (more than 4 weeks), or that could impact brain function at the time of the study. Subjects receiving psychotherapy may be included in the study.
6. Those with a binge drinking history every month continuously for the last 10 years will also be excluded. Binge drinkers are those who being female consume 4 or more drinks and males consume 5 or more drinks in one occasion at least once a month.
7. Serious neurological disorder such as MS, Parkinson s Disease, ALS, sensory loss or peripheral neuropathy.
8. Currently taking any psychoactive drugs such as Celexa (TM), Prozac (TM), Wellbutrin (TM), Zoloft (TM), and/or stimulants other than caffeine such as Adderall (TM), Dexedrine (TM) and Ritalin (TM). Subjects taking PRN medications (e.g., sleep medications) may be included in the study.
9. Clinically significant laboratory or examination results.
10. Study investigators and staff, as well as their superiors, subordinates and immediate family members (adult children, spouses, parents, siblings).
11. *Non-English speakers (must also be able to read and comprehend English).

    * The intent of the research has no prospect of direct benefit to the subject. Therefore, we are excluding non-English speakers in this research study since our fMRI paradigms (particularly the Delay Discounting task) require that the subject be able to speak, read and comprehend English.

Subjects will not be excluded from enrollment onto this study if their urine test or breath alcohol level (BAL) is positive for drugs/alcohol on initial screening. However, if they test positive on scheduled study procedure days involving MRI, the procedures will be postponed and rescheduled. We will allow for up to 3 rescheduled study days that were the result of positive urine drug or BAL screens. If the drug/BAL tests is/are positive on the third rescheduled visit, the participant will be withdrawn from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2016-06-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be amplitude and reliability of regional-specific BOLD fMRI signals. | end of study
  MRI: we will analyze measures such as the amplitude and the reliability of the test-retest measures of fMRI signals; functional connectivity metrics; tractography between seed and target regions of interest (diffusion tensor imaging, DTI); morphometry of brain regions (using automatic segmentation and voxel-brain morphometry, VBM); and brain metabolite levels in regions of interest (using MR spectroscopy, MRS).
The primary outcome will be amplitude and reliability of regional-specific BOLD fMRI signals. | end of study
  EEG (electroencephalography): we will quantify measures such as event or task-related potentials, and coherence between sensors or sources located close to the brain areas of interest. We are also quantifying blink rates from the electrooculogram (EOG).
The primary outcome will be amplitude and reliability of regional-specific BOLD fMRI signals. | end of study
  Behavioral measures during fMRI tasks: we will quantify measures such as reaction times and accuracy (using MRI compatible response pads) as well as eye movement (using MRI compatible eye trackers) and self-reports of the study experience (i.e. degree of interest and motivation and alertness).

SECONDARY OUTCOMES:
Collection of autonomic data | end of study
  Autonomic data may be collected or observations made during the course of the experiment that will give further information about the state of the body and emotions during experiments (blood pressure, skin conductance, respiratory rate). Self-report data may be collected during the course of the experiment to assess the level of interest, boredom, alertness of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Dardo G Tomasi, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The data will not be analyzed individually.

REFERENCES:
- [Background] Tomasi D, Wang GJ, Studentsova Y, Volkow ND. Dissecting Neural Responses to Temporal Prediction, Attention, and Memory: Effects of Reward Learning and Interoception on Time Perception. Cereb Cortex. 2015 Oct;25(10):3856-67. doi: 10.1093/cercor/bhu269. Epub 2014 Nov 11. PMID 25389123
- [Background] Tomasi D, Caparelli EC, Chang L, Ernst T. fMRI-acoustic noise alters brain activation during working memory tasks. Neuroimage. 2005 Aug 15;27(2):377-86. doi: 10.1016/j.neuroimage.2005.04.010. PMID 15893942
- [Background] Tomasi D, Wang R, Wang GJ, Volkow ND. Functional connectivity and brain activation: a synergistic approach. Cereb Cortex. 2014 Oct;24(10):2619-29. doi: 10.1093/cercor/bht119. Epub 2013 May 3. PMID 23645721
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-AA-0186.html